CLINICAL TRIAL: NCT06921551
Title: Exploratory Pilot Study on the Prolonged Use of the ABLE Exoskeleton in Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: Fundación Esclerosis Múltiple Madrid (FEMM) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABLEexoMSpost; CIV-24-10-049336 (Other: AEMPS)
Record Dates: First submitted 2025-03-27; First posted 2025-04-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Gait training; Wearable exoskeleton; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with exoskeleton (Experimental): Participants will undergo 60-min gait training sessions with the exoskeleton as part of their rehabilitation program once a week for up to 12 months
  Interventions: Device: ABLE Exoskeleton

INTERVENTIONS:
Device: ABLE Exoskeleton — Participants will undergo 60-min gait training sessions with the exoskeleton once a week for up to12 months

SUMMARY:
The goal of this study is to explore the potential clinical benefits of the ABLE Exoskeleton as part of a rehabilitation program in people with multiple sclerosis. The main question it aims to answer is:

Can a rehabiliation program with the ABLE Exoskeleton help to mantain the physical and psychosocial health of people with multiple sclerosis?

Participants will:

* Have a gait training session of 60 min with the exoskeleton once a week for 12 months at the clinic
* Have an evaluation (tests and questionnaires) every 3 months at the clinic

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* Diagnosed with multiple sclerosis
* Currently undergoing outpatient physical therapy treatment at the investigation site
* Ability to give informed consent

Exclusion Criteria:

* Significant osteoporosis that may increase the risk of fracture
* Unresolved fractures in the pelvis or extremities, or history of fragility fractures in the lower extremities in the last 2 years
* Spinal instability (or spinal orthoses, unless authorized by a physician)
* Severe spasticity: Level 4 on the Modified Ashworth Scale
* Orthostatic hypotension. Inability to tolerate a minimum of 30 minutes standing
* Uncontrolled autonomic dysreflexia
* Medical instability
* Unstable cardiovascular system (CVS), hemodynamic instability, untreated hypertension (SBP>140, DBP>90 mmHg), unresolved deep venous thrombosis (DVT)
* Serious comorbidities, including any condition that a physician deems inappropriate for use of the ABLE Exoskeleton or to complete participation in the study
* Skin integrity problems on the contact surfaces of the device or that would prevent sitting
* Grade I or higher on EPUAP (European Pressure Ulcer Advisory Panel, 2019) on areas that will be in contact with the exoskeleton
* Colostomy
* Anthropometric measurements outside the values compatible with ABLE Exoskeleton. In particular, height not between 1.5-1.9 m, or weight over 100 kg
* Anatomical constraints (such as eg length differences, users unable to position themselves inside the device) that are incompatible with the device
* Restrictions in range of motion that prevent normal gait from being achieved or preventing the completion of a normal transition from sitting to standing or standing to sitting
* Heterotopic ossification
* Known pregnancy or breastfeeding
* Cognitive impairment that results in the inability to follow simple instructions, particularly psychological or cognitive problems that do not allow a participant to follow study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Number of therapeutic objectives achieved | From baseline to the end of the training program at 12 months
  Two therapeutic objectives per participant will be defined at baseline. At the end of the training program, it will be assessed if the objectives were accomplished or not.
Lower extremity muscle strenght | Baseline, 3, 6, and 12 months post-training
  The Daniels Muscle Testing scale will be used to measure the strength of muscles in the lower extremities at baseline, every 3 months and at the end of the gait training program to assess motor function after the training. Scores range from 0 (absence of muscle activity) to 5 (normal muscle activity)
Modified Ashworth Scale (MAS) | Baseline, 3, 6, and 12 months post-training
  The Modified Ashworth Scale (MAS) measures spasticity in patients with lesions to the central nervous system. The scale assigns a grade of spasticity from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). It will be evaluated at baseline, every 3 months and at the end of the gait training program without the device to assess the change in the spasticity after training
Location and level of pain | Baseline, 3, 6, and 12 months post-training
  The location and level of pain using the numeric rating scale (NRS) will be assessed at baseline, every 3 months and at the end of the gait training program to assess the reduction of pain aftr the training
Timed 25-Feet Walk test (T25FW) | Baseline, 3, 6, and 12 months post-training
  The Timed 25-Foot Walk (T25FW) test measures the time a person needs to walk 25 feet. This test will be assessed at baseline, every 3 months, and at the end of the gait training program without the device to assess the change in the walking function after the training
6-Minute Walk Test (6MWT) | Baseline, 3, 6, and 12 months post-training
  The 6-Minute Walk Test (6MWT) measures the distance a person can walk in 6 minutes. This test will be assessed at baseline, every 3 months, and at the end of the gait training program without the device to assess the change in the walking function after the training
Borg Rating of Perceived Exertion | Baseline, 3, 6, and 12 months post-training
  The Borg Rating of Perceived Exertion (RPE) scale is used to measure a person's perception of their effort and exertion, breathlessness, and fatigue during physical activity. Scores range from 6 (no exertion at all) to 20 (maximal exertion). It will be evaluated during the 6MWT at baseline, every 3 months, and after the end of the gait training program without the device to assess the change in the perceived exertion after the training
Trunk Impairment Scale (TIS) | Baseline, 3, 6, and 12 months post-training
  The Trunk Impairment Scale (TIS) measures the motor impairment of the trunk through the evaluation of static and dynamic sitting balance as well as coordination of trunk movement. The total score ranges from 0 (minimal performance) to 23 (perfect performance). This test will be assessed at baseline, every 3 months, and at the end of the gait training program without the device to assess the change in the trunk impairment after training
Barthel Index (BI) score | Baseline, 3, 6, and 12 months post-training
  The Barthel Index (BI) will be used to assess the participants' ability to perform mobility and self-care activities of daily living (ADL). The total score ranges from 0 (total dependency) to 100 (independency). It will be evaluated at baseline, every 3 months, and after the gait training program without the device to assess the change in the independence to perform ADL after the training
Modified Fatigue Impact Scale (MFIS) score | Baseline, 3, 6, and 12 months post-training
  The Modified Fatigue Impact Scale (MFIS) provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning in persons with multiple sclerosis. The total score ranges from 0 to 84, with higher scores meaning a higher impact of fatigue. It will be evaluated iat baseline, every 3 months and at the end of the gait training program without the device to assess the change in the fatigue after the training
Multiple Sclerosis Quality of Life-54 (MSQoL-54) scores | Baseline, 3, 6, and 12 months post-training
  The Multiple Sclerosis Quality of Life-54 (MSQoL-54) is a multidimensional health-related quality of life (QoL) measure that combines both generic and MS-specific items into a single instrument. There is no single overall score for the MSQoL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores. The higher the score, the best the outcome. It will be evaluated at baseline, every 3 months and at the end of the gait training program without the device to assess the change in the QoL after the training
Self-perceived impact on general health status | 3, 6, and 12 months post-training
  Participants' perceptions of the impact on their general health will be evaluated by the completion of a self-report questionnaire on the perceived impact on general health. This questionnaire has been designed by the researchers and intends to identify to what extent participants feel that the ABLE Exoskeleton contributed to a change in their health. The questionnaire covers 7 categories (cardiovascular system, musculoskeletal pain, neuropathic pain, bladder and bowel, spasticity, and sleep quality) using a 7-point Likert scale to assess the change.
Level of motivation | After 12 months post-training
  Participants' perceptions on the level of motivation generated by the program with the ABLE Exoskeleton will be evaluated by the completion of a self-report questionnaire using a 7-point Likert scale. This questionnaire has been designed by the researchers.
Psychosocial Impact of Assistive Devices Scale (PIADS) score | After 12 months post-training
  The Psychosocial Impact of Assistive Devices Scale (PIADS) is a 26-item, self-reported questionnaire that provides a measure of user perception and other psychological factors associated with assistive technology devices. Scores range from -78 (maximum negative impact) to +78 (maximum positive impact). It will be used to assess the effects of the ABLE Exoskeleton on functional independence, well-being, and quality of life of participants after the training program experience
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) score | After 12 months post-training
  The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) is a 12-item outcome measure that assesses user satisfaction with two components (Device and Services) using a 5-point scale ranging from 1 (not satisfied) to 5 (very satisfied). Only the 8 items referred to the device will be evaluated from participants and the whole 12 items from the therapists to measure user satisfaction with the ABLE Exoskeleton after the training program experience

SECONDARY OUTCOMES:
Time spent upright and time spent walking | At session 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10
  In each gait training session, the time spent upright (in minutes) and the time spent walking (in minutes) with the device will be automatically measured and registered by the device
Number of steps walked | At session 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10
  In each gait training session, the number of steps taken (step count) with the device will be automatically measured and registered by the device
Distance walked | At session 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10
  In each gait training session, the distance walked (in meters) with the device will be automatically measured and registered by the device

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Esclerosis Múltiple Madrid (FEMM), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided